CLINICAL TRIAL: NCT00321230
Title: A Pilot Monocentric, Open Phase II Study to Investigate the Efficacy and Safety of a New Oral Gut Cleansing Solution ("Low Dose Bowel Prep") in 30 Patients Submitted to Colonoscopy
Brief Title: Clinical Evaluation of a New Reduced Volume Bowel Preparation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Marc Halphen, Norgine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRL994-02/2000; 02/2000
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Colonoscopy
Keywords: Colon cleansing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: macrogol3350 NA sulphate NACL KCL ascorbic acid NA ascorbate

SUMMARY:
Monocentric, cleansing evaluation pilot study in patients undergoing colonoscopy.

DETAILED DESCRIPTION:
Open prospective pilot monocentric phase II clinical trial evaluating the therapeutic efficacy of a new "Low Dose Bowel Prep" formulation for gut cleansing prior to colonoscopy.

Thirty patients admitted to the hospital (inpatients) planned to undergo a complete colonoscopy will have gut cleansing with the "Low Dose Bowel Prep" using a one-step intake mode.

ELIGIBILITY:
Inclusion Criteria:

* male or female, inpatients 18 to 65 years old with indication for complete colonoscopy
* the patient's written informed consent must be obtained prior to inclusion
* willing and able to complete the entire procedure and to comply with study instructions

Exclusion Criteria:

* ileus or toxic megacolon
* intestinal obstruction or perforation
* known of G6PD insufficiency
* history of any colonic surgery
* ischaemic cardiovascular disease
* untreated or uncontrolled arterial hypertension (max >170mmHg, min >100mmHg)
* renal insufficiency (creating above 45µmol/l)
* abnormal laboratory values (clinically significant) for sodium, potassium,chloride, creatinine and hematocrit
* cirrhosis of liver (Child-Pugh grade B or C)
* females who are pregnant, nursing or planning a pregnancy. Females of child bearing potential not using reliable methods of contraception.
* concurrent participation in an investigational drug study or participation within 30 days of study entry
* subject has a condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound the study results or may interfere significantly

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-01; Study Completion 2001-05

PRIMARY OUTCOMES:
Efficacy measured by a final scoring system i.e., "the overall quality of colonoscopy prep" that will be graded (from A to C) and assessed from the degree of cleansing in a 0 - 4 grade scale for each of the predefined colon areas.

SECONDARY OUTCOMES:
Stool weight as recorded on the case report form for each stool as from start of gut cleansing (day -1) to the beginning of colonoscopy (day 0).
Amount of fluid removed from the colon during the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Bitoun, MD, Principal Investigator — Hôpital Lariboisière
Locations (1):
- Hôpital Lariboisière, Endoscopy Department, Paris, France

REFERENCES:
- [Background] Davis GR, Santa Ana CA, Morawski SG, Fordtran JS. Development of a lavage solution associated with minimal water and electrolyte absorption or secretion. Gastroenterology. 1980 May;78(5 Pt 1):991-5. PMID 7380204